CLINICAL TRIAL: NCT01177111
Title: Impact of Sunflower Seed Oil Massage on Neonatal Mortality and Morbidity in Nepal
Acronym: NOMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Nepal Nutrition Intervention Project Sarlahi (Other); Tribhuvan University, Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD060712 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Neonatal Mortality; Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunflower seed Oil (Experimental)
  Interventions: Other: Sunflower seed oil
- Mustard seed oil (Active Comparator)
  Interventions: Other: Mustard seed oil

INTERVENTIONS:
Other: Sunflower seed oil — Locally manufactured refined sunflower seed oil will be provided to pregnant women late in pregnancy and community workers will promote its daily use during massage of newborns during the first month of life
  Arms: Sunflower seed Oil
Other: Mustard seed oil — Locally manufactured mustard seed oil will be provided to pregnant women late in pregnancy and community workers will promote its daily use during massage of newborns during the first month of life
  Arms: Mustard seed oil

SUMMARY:
Each year four million babies die during the neonatal period, with the majority occurring in developing countries. Overall, infections account for one-third of all neonatal deaths, with proportions approaching 50% in settings where neonatal mortality rates are high. Infections are predominately due to sepsis, respiratory infections, tetanus, and diarrhea. The investigators long term goal is to identify simple, affordable, and effective interventions that can be delivered at the community level in low-resource settings to reduce neonatal mortality risk due to these infections. The investigators team has conducted research in this area for the past 10 years, with specific focus on newborn vitamin A dosing and topical chlorhexidine antisepsis interventions. Previous community-based research by the investigators group of investigators and others demonstrated that newborn vitamin A dosing can reduce early infant mortality by approximately 20%, and that topical applications of chlorhexidine to the umbilical cord can prevent omphalitis and reduce neonatal mortality risk by 24%. Evidence is growing that neonatal skin plays an important role in protecting the newborn infant from invasive pathogens. Barrier function of the neonatal skin, however, is incomplete in newborn infants, especially those that are pre-term or of low birth weight. Full-body massage of newborns with mustard oil, practiced almost universally (~95%) in communities of south Asia, may further compromise skin barrier function through decreased structural integrity leading to increased trans-epidermal water loss and increased risk of percutaneous penetration by invasive pathogens. Loss of structural integrity is not seen after massage of neonatal skin with alternative topical emollients, including sunflower seed oil. Furthermore, sunflower seed oil has been shown to accelerate recovery of the skin barrier function, improve skin condition, and reduce the risk of both nosocomial infections and neonatal mortality among hospitalized newborns in low-resource settings. The specific hypothesis of this study is that substituting mustard oil with sunflower seed oil for topical applications during full body massage of newborns in the community will reduce neonatal mortality and morbidity by improving overall skin barrier function and reducing exposure to invasive pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Baby born alive
* Baby born in study area

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 29260 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
all cause neonatal mortality | first 28 days after birth
  A neonatal death is defined as death of a live born baby before completion of reaching 28.0 days old.
neonatal morbidity | first 28 days after birth
  Probable severe disease in newborns will be defined using the current World Health Organization (WHO) Young Infant Study Algorithm and appropriate adaptations

CONTACTS AND LOCATIONS:
Overall Officials: Luke C Mullany, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Nepal Nutrition Intervention Project, Hariaun, Sarlahi District, Nepal

REFERENCES:
- [Background] Thatte N, Mullany LC, Khatry SK, Katz J, Tielsch JM, Darmstadt GL. Traditional birth attendants in rural Nepal: knowledge, attitudes and practices about maternal and newborn health. Glob Public Health. 2009;4(6):600-17. doi: 10.1080/17441690802472406. PMID 19431006
- [Background] Falle TY, Mullany LC, Thatte N, Khatry SK, LeClerq SC, Darmstadt GL, Katz J, Tielsch JM. Potential role of traditional birth attendants in neonatal healthcare in rural southern Nepal. J Health Popul Nutr. 2009 Feb;27(1):53-61. doi: 10.3329/jhpn.v27i1.3317. PMID 19248648
- [Background] Mullany LC, Darmstadt GL, Khatry SK, Tielsch JM. Traditional massage of newborns in Nepal: implications for trials of improved practice. J Trop Pediatr. 2005 Apr;51(2):82-6. doi: 10.1093/tropej/fmh083. Epub 2005 Jan 26. PMID 15677372
- [Derived] Yue Y, Hazel EA, Subedi S, Zeger S, Mohan D, Mullany LC, Tielsch JM, Khatry SK, LeClerq SC, Katz J. Factors Predicting Completion of Four or More Antenatal Care Visits in Sarlahi District, Nepal. Res Sq [Preprint]. 2024 May 29:rs.3.rs-4467441. doi: 10.21203/rs.3.rs-4467441/v1. PMID 38853894
- [Derived] Katz J, Khatry SK, Shrestha L, Summers A, Visscher MO, Sherchand JB, Tielsch JM, Subedi S, LeClerq SC, Mullany LC. Impact of topical applications of sunflower seed oil on neonatal mortality and morbidity in southern Nepal: a community-based, cluster-randomised trial. BMJ Glob Health. 2024 Feb 29;9(2):e013691. doi: 10.1136/bmjgh-2023-013691. PMID 38423547
- [Derived] Yan T, Mullany LC, Subedi S, Hazel EA, Khatry SK, Mohan D, Zeger S, Tielsch JM, LeClerq SC, Katz J. Risk factors for neonatal mortality: an observational cohort study in Sarlahi district of rural southern Nepal. BMJ Open. 2023 Sep 14;13(9):e066931. doi: 10.1136/bmjopen-2022-066931. PMID 37709319
- [Derived] Subedi S, Hazel EA, Mohan D, Zeger S, Mullany LC, Tielsch JM, Khatry SK, LeClerq SC, Black RE, Katz J. Prevalence and predictors of spontaneous preterm births in Nepal: findings from a prospective, population-based pregnancy cohort in rural Nepal-a secondary data analysis. BMJ Open. 2022 Dec 1;12(12):e066934. doi: 10.1136/bmjopen-2022-066934. PMID 36456014
- [Derived] Hazel EA, Mohan D, Zeger S, Mullany LC, Tielsch JM, Khatry SK, Subedi S, LeClerq SC, Black RE, Katz J. Demographic, socio-economic, obstetric, and behavioral factors associated with small-and large-for-gestational-age from a prospective, population-based pregnancy cohort in rural Nepal: a secondary data analysis. BMC Pregnancy Childbirth. 2022 Aug 19;22(1):652. doi: 10.1186/s12884-022-04974-8. PMID 35986258
- [Derived] Subedi S, Katz J, Erchick DJ, Verhulst A, Khatry SK, Mullany LC, Tielsch JM, LeClerq SC, Christian P, West KP, Guillot M. Does higher early neonatal mortality in boys reverse over the neonatal period? A pooled analysis from three trials of Nepal. BMJ Open. 2022 May 19;12(5):e056112. doi: 10.1136/bmjopen-2021-056112. PMID 35589346
- [Derived] Erchick DJ, Khatry SK, Agrawal NK, Katz J, LeClerq SC, Rai B, Reynolds MA, Mullany LC. Risk of preterm birth associated with maternal gingival inflammation and oral hygiene behaviours in rural Nepal: a community-based, prospective cohort study. BMJ Open. 2020 Aug 20;10(8):e036515. doi: 10.1136/bmjopen-2019-036515. PMID 32819989
- [Derived] Erchick DJ, Agrawal NK, Khatry SK, Katz J, LeClerq SC, Rai B, Reynolds MA, Mullany LC. Feasibility of training community health workers to conduct periodontal examinations: a validation study in rural Nepal. BMC Health Serv Res. 2020 May 11;20(1):412. doi: 10.1186/s12913-020-05276-5. PMID 32393349
- [Derived] Summers A, Visscher MO, Khatry SK, Sherchand JB, LeClerq SC, Katz J, Tielsch JM, Mullany LC. Impact of sunflower seed oil versus mustard seed oil on skin barrier function in newborns: a community-based, cluster-randomized trial. BMC Pediatr. 2019 Dec 23;19(1):512. doi: 10.1186/s12887-019-1871-2. PMID 31870338
- [Derived] Erchick DJ, Rai B, Agrawal NK, Khatry SK, Katz J, LeClerq SC, Reynolds MA, Mullany LC. Oral hygiene, prevalence of gingivitis, and associated risk factors among pregnant women in Sarlahi District, Nepal. BMC Oral Health. 2019 Jan 5;19(1):2. doi: 10.1186/s12903-018-0681-5. PMID 30611255
- [Derived] Lubon AJ, Erchick DJ, Khatry SK, LeClerq SC, Agrawal NK, Reynolds MA, Katz J, Mullany LC. Oral health knowledge, behavior, and care seeking among pregnant and recently-delivered women in rural Nepal: a qualitative study. BMC Oral Health. 2018 Jun 1;18(1):97. doi: 10.1186/s12903-018-0564-9. PMID 29859084
- [Derived] Lama TP, Khatry SK, Katz J, LeClerq SC, Mullany LC. Illness recognition, decision-making, and care-seeking for maternal and newborn complications: a qualitative study in Sarlahi District, Nepal. J Health Popul Nutr. 2017 Dec 21;36(Suppl 1):45. doi: 10.1186/s41043-017-0123-z. PMID 29297386
- [Derived] Kozuki N, Katz J, Khatry SK, Tielsch JM, LeClerq SC, Mullany LC. Risk and burden of adverse intrapartum-related outcomes associated with non-cephalic and multiple birth in rural Nepal: a prospective cohort study. BMJ Open. 2017 Apr 20;7(4):e013099. doi: 10.1136/bmjopen-2016-013099. PMID 28428183